CLINICAL TRIAL: NCT00625703
Title: Pharmacokinetics of Linezolid in Children With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB File # 112007-010
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Cystic Fibrosis
Keywords: Pharmacokinetic
MeSH Terms: conditions — Cystic Fibrosis | interventions — Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Linezolid — Pharmacokinetics
  daily dose of linezolid at 15 mg/kg/dose Intravenously (IV) based on subject's weight at study entry, over half an hour period, every 8 hours for a minimum of 7 days to a maximum of 28 days total. The primary doctor may change the route of administration of linezolid from IV to oral (by mouth)after 72 hours on IV formulation and demonstrated clinical improvement based on the clinical evaluation by the primary doctor and comparison of cystic fibrosis exacerbation criteria scores before and after initiating treatment with linezolid.
  Other Names: Zyvox

SUMMARY:
To determine the pharmacokinetic profile of IV (intravenous) and PO (oral) formulations of linezolid among children with cystic fibrosis and establish a dose regimen that will be safe and effective.

DETAILED DESCRIPTION:
Patients with cystic fibrosis who have pulmonary exacerbations associated with the isolation of Methicillin-resistant Staphylococcus aureus (MRSA) in their sputum will be identified by their primary physicians and by laboratory record review. If they meet the inclusion criteria, they will be invited to participate in the study. The primary outcome variables include pharmacokinetic and pharmacodynamic indices. The study end points include completion of the sputum and blood sampling for pharmacokinetic studies of both intravenous and oral formulations of linezolid and collection of microbiologic specimen (sputum and anterior nares cultures) one month after discharge. Additionally, pharmacokinetic data will be analyzed for effects of age and cystic fibrosis transmembrane conductance regulator (CFTR) mutation on clearance of linezolid and for relationship between levels of linezolid achieved in sputum and blood and clinical outcome

ELIGIBILITY:
Inclusion Criteria:

* Subjects < 18 years of age inclusive, with a confirmed diagnosis of cystic fibrosis being admitted to the hospital for acute pulmonary exacerbation with MRSA isolated from sputum culture.
* Female subject of childbearing potential must have a negative pregnancy test prior to the first dose of study drug, and if sexually active agrees to use an acceptable method of birth control per investigator judgment for the duration of the study.
* Subjects who are receiving medications with serotonergic (such as certain types of antidepressants) and adrenergic activity that can not be discontinued based on clinical judgment of the primary physician may be enrolled. These subjects will be monitored closely for serotonin- and sympathomimetic-associated toxicity.
* Subject (when able) and subject's parent /legal guardian agree to comply with the study requirements.
* Subject has sufficient venous access to permit administration of the study medication, collection of pharmacokinetic samples and monitoring of safety variables.
* Duration of linezolid therapy is expected to exceed 7 days.
* English and Spanish-speaking subjects.

Exclusion Criteria:

* Subjects with clinical or laboratory evidence of severe hepatic (Child-Pugh class C) disease
* Subjects with severe renal impairment (estimated creatinine clearance <30 mL/min)
* Subjects with a history of allergy to linezolid.
* Pregnant and breastfeeding subjects.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2010-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Siegel, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No data available as PI is no longer at the institution. Several attempts were made to locate the PI or other study personnel associated with this study, but they were unsuccessful. Enrollment reflects the anticipated enrollment and actual enrollment is unknown due to PI is no longer at the institution.
Groups:
- Linezolid: Pharmacokinetics: daily dose of linezolid at 15 mg/kg/dose Intravenously (IV) based on subject's weight at study entry, over half an hour period, every 8 hours for a minimum of 7 days to a maximum of 28 days total. The primary doctor may change the route of administration of linezolid from IV to oral (by mouth)after 72 hours on IV formulation and demonstrated clinical improvement based on the clinical evaluation by the primary doctor and comparison of cystic fibrosis exacerbation criteria scores before and after initiating treatment with linezolid.
Period: Overall Study
Arm/Group | Linezolid: Pharmacokinetics
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No data available as PI is no longer at the institution. Several attempts were made to locate the PI or other study personnel associated with this study, but they were unsuccessful. Enrollment reflects the anticipated enrollment and actual enrollment is unknown due to PI is no longer at the institution.
Units Other Than Participants: participants
Arm/Group | Linezolid: Pharmacokinetics
Number analyzed (Participants) | 0
Number analyzed (participants) | 0
Age, Categorical
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Pharmacokinetic Profile of IV (Intravenous) and PO (Oral) Formulations of Linezolid Among Children With Cystic Fibrosis
Description: To determine the pharmacokinetic profile of IV (intravenous) and PO (oral) formulations of linezolid among children with cystic fibrosis and establish a dose regimen that will be safe and effective.
Time Frame: 2 months
Population: No data are available as PI is no longer at the institution. Several attempts were made to locate the PI or other study personnel associated with this study, but they were unsuccessful
Arm/Group | Linezolid: Pharmacokinetics
Number analyzed (Participants) | 0

2. Secondary Outcome: Pulmonary Exacerbations With Methicillin Resistant Staphylococcus Aureus (MRSA) to Treatment With Linezolid
Description: to characterize the clinical response of children with pulmonary exacerbations (increase in the severity of the patient's lung symptoms) associated with methicillin resistant Staphylococcus aureus (MRSA) to treatment with linezolid
Time Frame: 2 months
Population: as for outcome 1
Arm/Group | Linezolid: Pharmacokinetics
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: No data are available as PI is no longer at the institution. Several attempts were made to locate the PI or other study personnel associated with this study, but they were unsuccessful
Arm/Group | Linezolid: Pharmacokinetics
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linezolid: Pharmacokinetics (N=0)
Data not available (Investigations) | 0 (0) — No data are available as PI is no longer at the institution. Several attempts were made to locate the PI or other study personnel associated with this study, but they were unsuccessful
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linezolid: Pharmacokinetics (N=0)
No Data Available (Investigations) | 0 (0) — No data are available as PI is no longer at the institution. Several attempts were made to locate the PI or other study personnel associated with this study, but they were unsuccessful

LIMITATIONS AND CAVEATS:
No data are available as PI is no longer at the institution. Several attempts were made to locate the PI or other study personnel associated with this study, but they were unsuccessful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes